CLINICAL TRIAL: NCT01659203
Title: Phase I/II Trial of Pre-Operative Image Guided Intensity Modulated Proton Radiation Therapy (IMPT) or Photon (IMRT) With Simultaneously Integrated Boost to the High Risk Margin for Retroperitoneal Sarcomas
Brief Title: Proton or Photon RT for Retroperitoneal Sarcomas
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Roswell Park Cancer Institute (Other); National Cancer Institute (NCI) (NIH); Duke University (Other); Rush University Medical Center (Other); University of Utah (Other); Washington University School of Medicine (Other); Mayo Clinic (Other)
Responsible Party: Principal Investigator, Kevin X. Liu, MD, DPHIL, Radiation Oncologist, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-100
Record Dates: First submitted 2012-08-03; First posted 2012-08-07 (Estimated); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Retroperitoneal Sarcoma
Keywords: extraskeletal chondrosarcoma
MeSH Terms: conditions — Chondrosarcoma, Extraskeletal Myxoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment Arm IMPT (Experimental): IG-IMPT with SIB to the high risk margin
  Interventions: Radiation: IG-IMPT
- Treatment Arm IMRT (Experimental): IG IMRT with SIB to the high risk margin
  Interventions: Radiation: IG IMRT

INTERVENTIONS:
Radiation: IG-IMPT — Daily, Monday-Friday for about 6 weeks
  Arms: Treatment Arm IMPT
Radiation: IG IMRT — Daily, Monday-Friday for about 6 weeks
  Arms: Treatment Arm IMRT

SUMMARY:
This research study is a Phase I clinical trial. Phase I clinical trials test the safety of an investigational intervention. Phase I studies also try to define the appropriate dose of the investigational therapy to use for further studies. "Investigational" means that the intervention is still being studied and that research doctors are trying to find out more about it.

Retroperitoneal sarcomas are soft tissue tumors located at the far back of the abdomen. Typically, patients with retroperitoneal sarcomas either have surgery for the removal of their tumors alone, or have their tumors removed, followed by standard radiation therapy, or have pre-operative radiation followed by surgery. When conventional radiation therapy is delivered after surgery, it can damage normal tissue. In this study, you will undergo proton beam radiation therapy or IMRT before undergoing surgery for the removal of your tumor.

Proton radiation and IMRT are FDA approved radiation delivery systems. Protons are tiny particles with positive charge that can be controlled to travel a certain distance and stop inside the body. In theory, this allows better control of where the radiation dose is delivered as compared to photons. Since proton radiation is more targeted, it may help to reduce unwanted side effects from radiation.

In this study, a standard dose of radiation will be given to the majority of the tumor, while a simultaneously integrated boost of additional radiation will be given to certain areas of the tumor identified as higher risk. This means that a higher radiation dose will be given to the higher risk areas of the tumor.

The purpose of this study is to determine the highest dose of radiation therapy with protons or IMRT that can be delivered safely in patients with retroperitoneal sarcomas and the effectiveness of proton beam radiation therapy as an intervention for patients with retroperitoneal sarcomas.

DETAILED DESCRIPTION:
While being screened to determine eligibility for this study you may choose to participate in an additional blood sample for circulating DNA and a genomic DNA sample.

Since we are looking for the highest dose of Radiation Therapy that can be administered safely without severe or unmanageable side effects in participants that have retroperitoneal sarcomas, not everyone who participates in this research study will receive the same dose of study therapy. The dose you get will depend on the number of participants who have been enrolled in the study before you and how well they have tolerated their doses. Your study doctor will tell you which dose you will get.

Radiation planning is standard of care for all patients undergoing radiation therapy. Before you begin radiation therapy you will have a radiation planning CT scan of the tumor site. This scan will be in addition to the scans done in order to confirm your eligibility for this study. Doctors will use teh images from this scan to plan your radiation treatment.

You will receive radiation therapy every day Monday through Friday for about six weeks. You will receive study therapy as an outpatient. During radiation therapy, you will be seen by the study doctor once a week. Each visit will take about 15 minutes, and the following assessments will be completed: medical history, vital signs, body weight and assessments for any side effects you may be experiencing.

After the final dose of radiation therapy you will be assessed for side effects of radiation following your last dose and before surgery. The following assessments will be completed before your surgery at this visit: Chest CT, CT/MRI of the abdomen/pelvis and routine blood tests to check for overall health.

You will be seen for a follow-up visit within one month of discharge following surgery and again four months after the surgery. At the first follow-up visit, the following assessment will be completed: medical history, vital signs and body weight, questions about side effects and routine blood tests to check for overall health. At the four month follow up visit the following assessment will be completed: medical history, vital signs and body weight, chest CT and abdominal/pelvic CT.

After your four month follow-up visit, you will be seen twice yearly following radiation for the first five years and then once a year for the rest of your life.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven primary soft tissue sarcoma of the retroperitoneum
* Measurable disease
* Life expectancy of greater than 2 years

Exclusion Criteria:

* Prior radiation therapy for retroperitoneal sarcoma
* Pregnant or breastfeeding
* Chemotherapy within 4 weeks prior to entering study
* Receiving other investigational agents
* Other types of sarcomas
* Multifocal disease, lymph node or distant metastases
* History of sensitivity to radiation therapy
* Uncontrolled intercurrent illness
* History of a different invasive malignancy within the past 3 years
* HIV positive on combination anti-retroviral therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2012-12; Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Phase I: Determine MTD | 2 years
  To determine the maximum tolerated dose (MTD) of preoperative IG-IMPT or IMRTwith simultaneously integrated boost to the high risk margin of retroperitoneal sarcoma. This is mainly based on evaluation of acute toxicity profile of each participant.
Phase II: Determine Local Control Rate | 2 years
  To determine the local control rate after the protocol treatment (IG-IMPT or IMRT MTD with simultaneously integrated boost to the high risk margin) followed by surgical resection.

SECONDARY OUTCOMES:
Overall Survival | 2 years
  To estimate overall survival
Pathologic Response | 2 years
  To estimate pathologic response (percentage of necrosis and margin status, especially status of the high-risk margin)
Tumor Response | 2 years
  To estimate the tumor response through the comparison of CT imaging before and after the protocol treatment.
Progression-Free Survival Times | 2 years
  To assess progression-free survival times relative to surrogate biological endpoints in tissue and blood in each participant

CONTACTS AND LOCATIONS:
Overall Officials: Thomas F. DeLaney, M.D., Principal Investigator — Massachusetts General Hospital
Locations (10):
- United States (10):
  - Rush University Medical Center, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine Siteman Cancer Center West County, Creve Coeur, Missouri
  - Washington University School of Medicine Siteman Cancer Center South County, St Louis, Missouri
  - Roswell Park Cancer Institute, Buffalo, New York
  - Duke University, Durham, North Carolina
  - MD Anderson Cancer Center, Houston, Texas
  - University of Utah, Salt Lake City, Utah